CLINICAL TRIAL: NCT03686449
Title: Non-cultured Autologous Keratinocyte Suspension Versus Adipose-Derived Stem Cell-Keratinocyte Suspension for Coverage of Post-Burn Raw Area: A Comparative Clinical Study
Brief Title: Autologous Keratinocyte Suspension Versus Adipose-Derived Stem Cell-Keratinocyte Suspension for Post-Burn Raw Area
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Diefy Salem, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAKS-ADS
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Burn With Full-Thickness Skin Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- study group 1 (Experimental): Non-cultured Autologous Keratinocyte Suspension
  Interventions: Procedure: Non-cultured Autologous Keratinocyte Suspension
- study group 2 (Experimental): Adipose-Derived Stem cell-Keratinocyte Suspension
  Interventions: Procedure: Adipose-Derived Stem cell-Keratinocyte Suspension
- Control group (Active Comparator): Split skin graft
  Interventions: Procedure: Split skin graft

INTERVENTIONS:
Procedure: Non-cultured Autologous Keratinocyte Suspension — New method for treatment of post-burn raw area
  Arms: study group 1
Procedure: Adipose-Derived Stem cell-Keratinocyte Suspension — New method for treatment of post-burn raw area
  Arms: study group 2
Procedure: Split skin graft — Traditional method for treatment of post-burn raw area
  Arms: Control group

SUMMARY:
In this study

1. Assess the efficiency of non-cultured autologous keratinocyte suspension in treating post-burn raw area.
2. Compare the results of keratinocyte suspension alone versus Adipose-derived mesenchymal stem cells-keratinocyte suspension in post-burn raw area.

DETAILED DESCRIPTION:
Burn injuries are complicated wounds to manage with a relative high mortality rate in especially large area burns and elderly patients.

Substantial tissue damage and extensive fluid loss can cause impaired vital functions of the skin. When healing is delayed, the potential short term common complications include wound infection affecting the local healing process or systemic inflammatory and immunological responses which subsequently can cause life threatening sepsis and multi-organ failure.

Fortunately, survival rates have improved drastically over the last century due to advancements in burn care such as early surgical intervention, critical care support and wound care.

For many years the "gold standard" for treating wounds of burn patients has been transplantation with an autologous split skin graft. In patients with extensive burn wounds donor sites may be limited. In order to cover all the wounds, the patients often need multiple operations and/or the skin had to be expanded as much as possible.

However, the current different expansion techniques and treatments [mesh and Meek-Wall] frequently lead to scar formation, especially in the large mesh intersites.

The rate of wound closure depends on how quickly epidermal cells migrate out of the meshed auto graft and/ or wound edges to close the wound. Accelerating re-epithelialization could potentially improve the outcome of the healing process in terms of reducing granulation tissue formation, reducing the healing time, and thereby reducing the risk of colonization and infection, as well as scar formation.

Since clinical cases were first successfully treated with cultured epithelial layers, keratinocyte sheets have become an important tool in burn wound treatment. However, the clinical application can be limited by long culture time and fragility of the keratinocyte sheets. There is, therefore, a clinical demand for other options to cover large areas of burn wounds in the absence of viable donor sites.

A novel concept consists of treating wounds with epithelial cell suspensions. In 1998, Fraulin et al. developed a method of spreading cell suspension on to wounds using an aerosol spray in a porcine model.

The use of non-cultured keratinocyte suspensions was first reported by Hunyadi et al., showing that a group of patients with burn wounds or chronic leg ulcers, treated with a fibrin matrix containing keratinocytes, healed completely, as opposed to the control group.

In porcine wound models, non-cultured keratinocyte suspensions have been shown to accelerate wound healing, improve quality of epithelialization, and restore melanocyte population, compared to the respective control group.

Major advantages in the use of non-cultured cell suspensions are a drastic reduction of preparation time and possibly easier handling compared to keratinocyte sheets. Particularly, scar quality may be improved by enhancing the speed of epithelialization and fading of mesh patterns in split skin grafts.

On the other hand, stem cell-based therapies have gained interest as a promising approach to enhance tissue regeneration.

Stem cells are characterized by their multipotency and capacity for self-renewal. Their therapeutic potential is largely due to their ability to secrete proregenerative cytokines, making them an attractive option for the treatment of chronic wounds.

Stem cells from numerous sources are currently being tested in preclinical and clinical trials for their ability to faster wound healing and tissue regeneration. These trials have not only proven autologous stem cell therapy to be safely tolerated, but also demonstrated positive clinical outcomes.

According to the International Society of Cellular Therapy, mesenchymal stem cells are defined by their ability to adhere to a plastic surface, by their expression of the surface markers CD73, CD90, and CD105, by their lack of expression of hematopoietic markers CD14, CD34, CD45, CD11b/CD79, and CD19/HLA-DR, and by their ability to differentiate along osteoblastic, adipocytic and chondrocytic pathways.

Isolated from tissues including bone marrow, adipose tissue, umbilical cord blood, nerve tissue, and dermis, MSCs have been administered both systemically and locally for the treatment of cutaneous wounds.18 Although mesenchymal stem cells have been shown to exhibit low levels of long-term incorporation into healing wounds, a growing body of research suggests that their therapeutic benefit is attributed to their release of trophic mediators, rather than a direct structural contribution.19 Through the release of vascular endothelial growth factor, stromal cell-derived factor-1, epidermal growth factor, keratinocyte growth factor, insulin-like growth factor, and matrix metalloproteinase-9, mesenchymal stem cells promote new vessel formation, recruit endogenous progenitor cells, and direct cell differentiation, proliferation, and extracellular matrix formation during wound repair.

Mesenchymal stem cells also exhibit key immunomodulatory properties though the secretion of interferon-λ, tumor necrosis factor-α, interleukin-1α and interleukin-1β, as well as through the activation of inducible nitric oxide synthase. Mesenchymal stem cells secretion of prostaglandin E2 further regulates fibrosis and inflammation, promoting tissue healing with reduced scarring.

Finally, Mesenchymal stem cells display bactericidal properties through the secretion of antimicrobial factors and by upregulating bacterial killing and phagocytosis by immune cells.

Adipose-derived mesenchymal stem cells are a pluripotent, heterogeneous population of cells present within human adipose tissue.

However, isolation of adipose-derived mesenchymal stem cells is readily accomplished using liposuction aspirates or excised fat samples, which are obtainable with minimal donor morbidity.

Adipose-derived mesenchymal stem cells can be differentiated into adipogenic, chondrogenic, myogenic, and osteogenic cell lineages in response to specific stimuli. Alternatively, adipose-derived mesenchymal stem cells may be immediately administered without in vitro expansion or differentiation in culture.

The extraordinarily high cell yield from lipoaspirate (as many as 1*107 cells from 300 ml of lipoaspirate with at least 95% purity), as compared with bone marrow aspiration, makes Adipose-derived mesenchymal stem cells a particularly attractive cell source for the acute wound setting.

ELIGIBILITY:
Inclusion Criteria:

* Post-burn raw area more than 10% total body surface area

Exclusion Criteria:

* Presence of pre-existing local and systemic bacterial infections.
* Pre-existing medical conditions that would interfere with wound healing (i.e. uncontrolled diabetes mellitus, malignancy, congestive heart failure, autoimmune disease, renal failure, corticosteroids and immunosuppressive drugs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Length of the operating procedure | 1 day

SECONDARY OUTCOMES:
The mean time to 95% healing of the burn wound | 1 month

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jackson PC, Hardwicke J, Bamford A, Nightingale P, Wilson Y, Papini R, Moiemen N. Revised estimates of mortality from the Birmingham Burn Centre, 2001-2010: a continuing analysis over 65 years. Ann Surg. 2014 May;259(5):979-84. doi: 10.1097/SLA.0b013e31829160ca. PMID 23598383
- [Background] Osler T, Glance LG, Hosmer DW. Simplified estimates of the probability of death after burn injuries: extending and updating the baux score. J Trauma. 2010 Mar;68(3):690-7. doi: 10.1097/TA.0b013e3181c453b3. PMID 20038856
- [Background] Deitch EA, Wheelahan TM, Rose MP, Clothier J, Cotter J. Hypertrophic burn scars: analysis of variables. J Trauma. 1983 Oct;23(10):895-8. PMID 6632013
- [Background] Hefton JM, Madden MR, Finkelstein JL, Shires GT. Grafting of burn patients with allografts of cultured epidermal cells. Lancet. 1983 Aug 20;2(8347):428-30. doi: 10.1016/s0140-6736(83)90392-6. PMID 6135914
- [Background] Fraulin FO, Bahoric A, Harrop AR, Hiruki T, Clarke HM. Autotransplantation of epithelial cells in the pig via an aerosol vehicle. J Burn Care Rehabil. 1998 Jul-Aug;19(4):337-45. doi: 10.1097/00004630-199807000-00012. PMID 9710733
- [Background] Hunyadi J, Farkas B, Bertenyi C, Olah J, Dobozy A. Keratinocyte grafting: a new means of transplantation for full-thickness wounds. J Dermatol Surg Oncol. 1988 Jan;14(1):75-8. doi: 10.1111/j.1524-4725.1988.tb03343.x. PMID 2447135
- [Background] Behr B, Ko SH, Wong VW, Gurtner GC, Longaker MT. Stem cells. Plast Reconstr Surg. 2010 Oct;126(4):1163-1171. doi: 10.1097/PRS.0b013e3181ea42bb. PMID 20555302
- [Background] Garg RK, Rennert RC, Duscher D, Sorkin M, Kosaraju R, Auerbach LJ, Lennon J, Chung MT, Paik K, Nimpf J, Rajadas J, Longaker MT, Gurtner GC. Capillary force seeding of hydrogels for adipose-derived stem cell delivery in wounds. Stem Cells Transl Med. 2014 Sep;3(9):1079-89. doi: 10.5966/sctm.2014-0007. Epub 2014 Jul 18. PMID 25038246
- [Background] Kirana S, Stratmann B, Prante C, Prohaska W, Koerperich H, Lammers D, Gastens MH, Quast T, Negrean M, Stirban OA, Nandrean SG, Gotting C, Minartz P, Kleesiek K, Tschoepe D. Autologous stem cell therapy in the treatment of limb ischaemia induced chronic tissue ulcers of diabetic foot patients. Int J Clin Pract. 2012 Apr;66(4):384-93. doi: 10.1111/j.1742-1241.2011.02886.x. Epub 2012 Jan 27. PMID 22284892
- [Background] Caplan AI, Dennis JE. Mesenchymal stem cells as trophic mediators. J Cell Biochem. 2006 Aug 1;98(5):1076-84. doi: 10.1002/jcb.20886. PMID 16619257
- [Background] Badiavas EV, Falanga V. Treatment of chronic wounds with bone marrow-derived cells. Arch Dermatol. 2003 Apr;139(4):510-6. doi: 10.1001/archderm.139.4.510. PMID 12707099
- [Background] Hu MS, Rennert RC, McArdle A, Chung MT, Walmsley GG, Longaker MT, Lorenz HP. The Role of Stem Cells During Scarless Skin Wound Healing. Adv Wound Care (New Rochelle). 2014 Apr 1;3(4):304-314. doi: 10.1089/wound.2013.0471. PMID 24761362
- [Background] Zuk PA, Zhu M, Ashjian P, De Ugarte DA, Huang JI, Mizuno H, Alfonso ZC, Fraser JK, Benhaim P, Hedrick MH. Human adipose tissue is a source of multipotent stem cells. Mol Biol Cell. 2002 Dec;13(12):4279-95. doi: 10.1091/mbc.e02-02-0105. PMID 12475952
- [Background] Boquest AC, Shahdadfar A, Brinchmann JE, Collas P. Isolation of stromal stem cells from human adipose tissue. Methods Mol Biol. 2006;325:35-46. doi: 10.1385/1-59745-005-7:35. PMID 16761717